CLINICAL TRIAL: NCT00442780
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose Escalation Study of Multiple Doses of BIIB014 Administered Orally in Subjects With Early Parkinson's Disease
Brief Title: Dose-Finding Safety Study of BIIB014 in Early-Stage Parkinson's Disease
Acronym: MOBILE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Biogen Idec MD, Biogen Idec
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 204PD203; EUDRA CT NO: 2007-000398-47
Record Dates: First submitted 2007-03-01; First posted 2007-03-02 (Estimated); Last update posted 2009-01-09 (Estimated); Status verified 2009-01

CONDITIONS: Parkinson's Disease
Keywords: early Parkinson's Disease; MOBILE; BIIB014
MeSH Terms: conditions — Parkinson Disease | interventions — 3-(4-amino-3-methylbenzyl)-7-(2-furyl)-3H-(1,2,3)triazolo(4,5-d)pyrimidine-5-amine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Placebo Comparator): Dose Level A of BIIB014
  Interventions: Drug: BIIB014; Drug: Placebo
- 2 (Placebo Comparator): Dose Level B of BIIB014
  Interventions: Drug: BIIB014; Drug: Placebo
- 3 (Placebo Comparator): Dose Level C of BIIB014
  Interventions: Drug: BIIB014; Drug: Placebo
- 4 (Placebo Comparator): Dose Level D of BIIB014
  Interventions: Drug: BIIB014; Drug: Placebo

INTERVENTIONS:
Drug: BIIB014 — oral administration of BIIB014 per dose, schedule,and duration specified in protocol
Drug: Placebo — Oral administration of placebo matched to BIIB014 dose level; placebo to follow same dosing schedule as BIIB014

SUMMARY:
The main purpose of this study is to determine the safety of BIIB014 and how well BIIB014 is tolerated when given at different doses to patients with early-stage Parkinson's Disease.

This study will also explore:

* How BIIB014 is affected when given to patients with early-stage Parkinson's Disease (this will be done by measuring the levels of BIIB014 in the blood at several different times during the study), and
* The activity of BIIB014 when given to early Parkinson's patients (this will be done by performing different Parkinson's Disease assessments and other tests during the study).

Patients who enter this study will be randomly assigned to receive either BIIB014 or a placebo but because the study is blinded, neither they nor their study doctor will know which study treatment they are taking.

ELIGIBILITY:
Inclusion Criteria:

* Must give written informed consent and any authorizations required by local law.
* Must carry a diagnosis of idiopathic Parkinson's Disease(PD), without any other known or suspected cause of parkinsonism, according to the UK Parkinson's Disease Society Brain Bank Clinical Diagnostic Criteria. Initial diagnosis of PD must have been made within the 5 years prior to Screening with at least two or more of the following cardinal signs being present: bradykinesia, resting tremor, rigidity, and postural instability.
* Must be modified Hoehn & Yahr Stage 1 to 2.5 (inclusive).
* Must have a baseline UPDRS (Part III) motor score of at least 10.
* Subjects may be receiving an anticholinergic agent and/or MAO-B inhibitor (if they have been on a stable dose of that medication for at least 4 weeks prior to study entry) but must not be receiving any other PD medication.

Exclusion Criteria:

* A Mini Mental State Examination (MMSE) score <26.
* History or clinical features consistent with an atypical parkinsonian syndrome.
* Any significant non-PD central nervous system disorder.
* Any significant AXIS I psychiatric disease as defined by the Diagnostic and Statistical Manual of Mental Disorders.
* History of cognitive or neuropsychiatric conditions.
* History of surgical intervention for PD.
* History of L-DOPA-induced motor or non-motor complication.
* History of malignancy.
* History of severe allergic or anaphylactic reactions to any drug.
* Clinically significant renal dysfunction.
* HbA1c >7.0%.
* Clinically significant baseline ECG.
* Orthostatic hypotension.
* Treatment with L-DOPA/carbidopa or L-DOPA/benserazide for more than 6 cumulative months at anytime since subject's initial PD diagnosis.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2007-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Number and proportion of subjects with adverse events | up to end of study
Assessment of clinical laboratory parameters. | up to end of study
Assessment of vital signs. | up to end of study
Assessment of ECG parameters. | up to end of study

SECONDARY OUTCOMES:
Assess PK by measuring concentrations of BIIB014 and its N-acetyl metabolite in blood plasma. | up to end of study
Explore BIIB014 activity by evaluating standard Parkinson's disease assessments. | up to end of study
Explore the PK/pharmacodynamic relationships for BIIB014. | up to end of study

CONTACTS AND LOCATIONS:
Overall Officials: Biogen Idec, MD, Study Director — Cambridge, MA USA
Locations (10):
- Israel (4):
  - Research Site, Ashkelon
  - Research Site, Petah Tikva
  - Research Site, Ramat Gan
  - Research Site, Tel Aviv
- Poland (4):
  - Research Site, Kielce
  - Research Site, Krakow
  - Research Site, Poznan
  - Research Site, Warsaw
- Serbia (2):
  - Research Sites, Belgrade
  - Research Site, Belgrade